CLINICAL TRIAL: NCT00313690
Title: Phase I/II Study of Neoadjuvant Bortezomib in Combination With Docetaxel and Cisplatin Followed by Surgery in Early Stage Non-Small Cell Lung Cancer.
Brief Title: Cancer Treatment Followed by Surgery for Early Stage Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Southern California (Other)
Responsible Party: Barbara Gitlitz, MD, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2N-05-2
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bortezomib; Docetaxel; Cisplatin

INTERVENTIONS:
Drug: Bortezomib, Docetaxel and Cisplatin

SUMMARY:
* The purpose of the phase I portion of the study is to determine the safety and feasibility of neoadjuvant bortezomib in combination with docetaxel and cisplatin followed by surgery in early stage non-small cell lung cancer, via a multi-cohort dose escalation trial.
* The phase II portion of the study will look at the clinical response rate and the pathology response rate. Other purposes are to look at surgical morbidity, mortality and respectability rates. Molecular correlates of response and survival to this neoadjuvant regimen will be explored.

ELIGIBILITY:
Inclusion Criteria:(Phase I and II unless otherwise specified)

* Potential subjects may either be suspected to have non-small cell lung cancer with plans for a diagnostic biopsy, or must have a histological or cytological diagnosis of non-small cell lung cancer. For those suspected of having non-small cell lung cancer, histological confirmation must be obtained prior to commencing treatment on protocol. During the phase II portion of this protocol, all subjects will be asked to undergo FNA/core biopsy of the primary tumor for correlative studies even if they already came to screening with prior biopsy (histological confirmation of disease). However, subjects refusing repeat FNA/core biopsy will not be excluded from protocol entry
* Subjects must have stage IB ,IIA ,or IIIA. T stage must be defined by CT and PET imaging. Nodal status must be determined by CT/PET imaging, N2 disease must be confirmed by mandatory mediastinoscopy
* Subjects must be chemotherapy and radiation therapy naïve
* No history of prior malignancy except adequately treated basal cell or squamous cell skin cancer, or adequately treated cervical carcinoma in situ.
* Age greater than 18 years.
* Zubrod performance status of 0 or 1.
* Patients must have adequate organ and marrow function as defined below:
* absolute neutrophil count greater than or equal to 1,500
* platelets greater than or equal to 100,000/ml
* total bilirubin within normal institutional limits
* hemoglobin greater than 8.0 g/dl
* AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility.
* Creatinine within normal institutional limits OR Calculated creatinine clearance greater than or equal to 60 ml/min.
* Female subject of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry, during treatment and for at least 3 months thereafter. Women of child bearing potential must have a documented negative pregnancy associated ß-HCG during screening.
* Predicted post-resection FEV1 of 1.0 L or more
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects must not be receiving nor plan on receiving any other investigational agents.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* History of known allergy to compounds of similar chemical or biologic composition to bortezomib or other agents used in this study (i.e. Boron, Mannitol).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, congestive heart failure or myocardial infarction within the preceding 6 months, symptomatic cardiac arrhythmia, unstable angina pectoris, psychiatric illness or social situations that would limit compliance with study prescribed therapy.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients are excluded from the study.
* Pregnant or nursing women
* Peripheral neuropathy: greater than grade 1
* Inclusion of Women and Minorities

Both men and women of all ethnic groups are eligible for this trial if they meet the eligibility criteria. To date, there is no information that suggests differences in drug metabolism or disease response would be expected in one group compared to another. All efforts will be made to accrue a representative sample. If differences in outcome appear to be associated with gender or ethnicity, then perhaps a follow-up study can be designed to investigate these differences more fully. The catchment's area for USC is Los Angeles County.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, MD, Principal Investigator — USC Comprehensive Cancer Center